CLINICAL TRIAL: NCT05126407
Title: A Non-Interventional Clinical Study to Assess the Risk and Performance Aspects of Olynth Saline/Ectomed Nasal Drops/Spray Based Upon Previous Usage
Brief Title: A Study of Olynth Saline/Ectomed Nasal Drops/Spray Based Upon Previous Usage
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Other Study IDs: CCSURA003229; CCSURA003229 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-11-03; First posted 2021-11-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Common Cold; Sinusitis; Hypersensitivity
MeSH Terms: conditions — Common Cold; Sinusitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Olynth Nasal Saline Drops/Spray and Olynth Ectomed Nasal Spray: Participants who have personally used or administered the Olynth Nasal Saline Drops/Spray and Olynth Ectomed Nasal Spray to a child at least once within the past 6 months will provide feedback via electronic survey on the prior use of the Drop/Spray.

SUMMARY:
The purpose of this study is to proactively collect customer feedback on the performance aspects and risk factors of Olynth Nasal Saline Drops/Spray and Olynth Ectomed Nasal Spray.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older who has personally used or administered the nasal drops/spray to a child
* Has personally used or administered to a child, the Nasal Drops/Spray at least once within the past 6 months
* Able to read, write, speak, and understand German
* Has internet access to complete an on-line survey
* Intends to complete the survey
* Individual has signed the informed consent document (ICD)

Exclusion Criteria:

- Is an employee/contractor or immediate family member of the principal investigator (PI), Schlesinger group, product perceptions limited (PPL) Insights or sponsor of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who has personally used or administered the Olynth Nasal Saline Drops/Spray and Olynth Ectomed Nasal Spray to a child will be included.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Participant Feedback on the Performance Aspects of Olynth Nasal Saline Drops | Up to 1 month and 14 days
  Participant feedback on the performance aspects of Olynth Nasal Saline Drops will be assessed via electronic survey.
Participant Feedback on the Performance Aspects of Olynth Nasal Saline Spray | Up to 1 month and 14 days
  Participant feedback on the performance aspects of Olynth Nasal Saline Spray will be assessed via electronic survey.
Participant Feedback on the Performance Aspects of Olynth Ectomed Nasal Spray | Up to 1 month and 14 days
  Participant feedback on the performance aspects of Olynth Ectomed Nasal Spray will be assessed via electronic survey.
Number of Participants with Adverse Events (AEs) | Up to 1 month and 14 days
  An AE is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, including an abnormal laboratory finding, in participants, users or other persons, whether or not related to the investigational device.

CONTACTS AND LOCATIONS:
Overall Officials: Akash Pandhare, MD. Ph.D., Principal Investigator — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- Schlesinger Group, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Spector SL, Toshener D, Gay I, Rosenman E. Beneficial effects of propylene and polyethylene glycol and saline in the treatment of perennial rhinitis. Clin Allergy. 1982 Mar;12(2):187-96. doi: 10.1111/j.1365-2222.1982.tb01638.x. PMID 7074822
- [Background] Chirico G, Quartarone G, Mallefet P. Nasal congestion in infants and children: a literature review on efficacy and safety of non-pharmacological treatments. Minerva Pediatr. 2014 Dec;66(6):549-57. PMID 25336097
- [Background] Eichel A, Wittig J, Shah-Hosseini K, Mosges R. A prospective, controlled study of SNS01 (ectoine nasal spray) compared to BNO-101 (phytotherapeutic dragees) in patients with acute rhinosinusitis. Curr Med Res Opin. 2013 Jul;29(7):739-46. doi: 10.1185/03007995.2013.800474. Epub 2013 May 14. PMID 23621514
- [Background] Koksal T, Cizmeci MN, Bozkaya D, Kanburoglu MK, Sahin S, Tas T, Yuksel CN, Tatli MM. Comparison between the use of saline and seawater for nasal obstruction in children under 2 years of age with acute upper respiratory infection. Turk J Med Sci. 2016 Jun 23;46(4):1004-13. doi: 10.3906/sag-1507-18. PMID 27513397
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSURA003229&attachmentIdentifier=c0fde2b4-7ed1-4748-9c55-a00844306b24&fileName=256062_Project_Rudolph_Final_Synopsis16JUN2022_.pdf&versionIdentifier=